CLINICAL TRIAL: NCT06187441
Title: FeAsiBility of a Treatment Free Interval in Newly Diagnosed mUltiple myeLOma Patients Treated With DaratumUmab-Lenalidomide-DexamethaSone- the FABULOUS Study. A Nationwide Open-label Randomized Phase III Clinical Trial Comparing Daratumumab-lenalidomide-dexamethasone Continuously Versus Including a Treatment Free Interval
Brief Title: FeAsiBility of a Treatment Free Interval in Newly Diagnosed MM Patients Treated With Daratumumab-lenalidomide-dexamethasone (HOVON174MM)
Acronym: HOVON174MM
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stichting Hemato-Oncologie voor Volwassenen Nederland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HO174; 2023-508586-33-00 (Other: EU CT)
Record Dates: First submitted 2023-12-01; First posted 2024-01-02 (Actual); Last update posted 2024-08-19 (Actual); Status verified 2024-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — daratumumab; Dexamethasone; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (No Intervention): A continuous therapy arm - continuation of therapy with Dara-Rd until PD
- Arm B (Experimental): treatment free interval arm - discontinuation of therapy with Dara-Rd, which will be resumed at biochemical progression and given until PD
  Interventions: Drug: Daratumumab Injection; Drug: Dexamethasone; Drug: Lenalidomide capsule

INTERVENTIONS:
Drug: Daratumumab Injection — Patients who have been treated with 12 cycles of Daratumumab-Lenalidomide-Dexamethasone (Dara-Rd) will be randomized between Arm A (continuous therapy) and Arm B (treatment free interval)
  Arms: Arm B
Drug: Dexamethasone — Patients who have been treated with 12 cycles of Daratumumab-Lenalidomide-Dexamethasone (Dara-Rd) will be randomized between Arm A (continuous therapy) and Arm B (treatment free interval)
  Arms: Arm B
Drug: Lenalidomide capsule — Patients who have been treated with 12 cycles of Daratumumab-Lenalidomide-Dexamethasone (Dara-Rd) will be randomized between Arm A (continuous therapy) and Arm B (treatment free interval)
  Arms: Arm B

SUMMARY:
In the Netherlands, the standard treatment for multiple myeloma is a combination of different medicines named daratumumab-lenalidomide-dexamethasone, abbreviated as Dara-Rd. In many patients this treatment results in suppressing the disease for a long time. The treatment is continued until it is not effective anymore and the disease progresses.

But until now it is unknown whether continuous therapy also leads to prolonging life. In addition, there are concerns about side effects, leading to a reduced quality of life, the development of severe toxicity that remains, which hampers subsequent therapy, and high costs due to prolonged treatment.

There are indications that temporarily stopping treatment is safe, leading to fewer side effects and allows recovering from toxicity or damage due to treatment. This may improve the quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Patient was diagnosed with MM, based on the IMWG criteria, and measurable disease at the time of diagnosis (appendix A).
* Age ≥ 18 years.
* Patient was treated with 12 cycles (13 cycles is accepted) of Dara-Rd and will continue treatment with Dara-Rd. Reduced dosing of lenalidomide, but not to less than 5 mg, and previous discontinuation or dose reduction of dexamethasone is allowed.
* Partial response or better after treatment with 12 cycles of Dara-Rd, without signs of biochemical progression.
* ANC ≥ 1.0x109/L and platelets ≥ 75x109/L.
* Patient is capable of giving informed consent.
* Written informed consent.

Exclusion Criteria:

* Patient with non-secretory MM at diagnosis of the disease, i.e., before the start of treatment with Dara-Rd.
* Patient in whom a plasmacytoma was the only measurable parameter at diagnosis of the disease, i.e., before the start of treatment with Dara-Rd.
* Patient in whom urine M-protein was the only measurable parameter at diagnosis of the disease, i.e., before the start of treatment with Dara-Rd.
* Patient in whom treatment with daratumumab, lenalidomide or both has been discontinued for whatever reason (patients may only have discontinued dexamethasone).
* Patient in whom continuation of treatment with Dara-Rd is deemed not feasible because of medical reasons.
* Any psychological, familial, sociological and geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 599 (Estimated)
Dates: Start 2024-05-14 (Actual); Primary Completion 2031-01 (Estimated); Study Completion 2037-12 (Estimated)

PRIMARY OUTCOMES:
Compare Event-Free Survival (EFS) | Approximately up to 57 (EFS) months after randomization of the first patient
  To compare Event-Free Survival (EFS) from the time of randomization, between arm A continuous therapy with Dara-Rd until PD versus arm B discontinuation of therapy with Dara-Rd, resuming therapy at the first signs of biochemical progression until PD
Compare Progression Free Survival (PFS) | Approximately up to 69 (PFS) months after randomization of the first patient
  To compare Progression Free Survival (PFS) from the time of randomization, between arm A continuous therapy with Dara-Rd until PD versus arm B discontinuation of therapy with Dara-Rd, resuming therapy at the first signs of biochemical progression until PD

SECONDARY OUTCOMES:
Compare adverse event burden | Approximately up to 69 months after randomization of the first patient
  To compare adverse event (AE) burden between arms
Compare patient-reported outcome measures (PROMs) | Approximately up to 69 months after randomization of the first patient
  To compare PROMs between arms via validated questionnaires such as Impact of Cancer version 2 Cancer Worry scale
Compare cost-effectiveness between arms | Approximately up to 69 months after randomization of the first patient
  To compare cost-effectiveness between arms
Determine the length of the treatment-free interval | Approximately up to 69 months after randomization of the first patient
  To determine the length of the treatment-free interval (TFI) in arm B
Determine time to (maximal) response response | Approximately up to 69 months after randomization of the first patient
  To determine time to (maximal) response after restart of Dara-Rd in arm B.
Compare time to next treatment | Approximately up to 69 months after randomization of the first patient
  To compare time to next treatment (TTNT) between arms
Compare time from randomization to progression on second-line therapy | Approximately up to 69 months after randomization of the first patient
  To compare time from randomization to progression on second-line therapy (PFS2) between arms.
Compare Overall Survival | Approximately up to 69 months after randomization of the last patient
  To compare Overall Survival (OS) between arms.
Compare the discontinuation rate | Approximately up to 69 months after randomization of the first patient
  To compare the discontinuation rate and the reasons for discontinuation between arms.
Evaluate cumulative doses | Approximately up to 69 months after randomization of the first patient
  To evaluate cumulative dose of daratumumab, lenalidomide and dexamethasone in both arms.
Compare dose reductions | Approximately up to 69 months after randomization of the first patient
  To compare dose reductions of daratumumab, lenalidomide and dexamethasone between arms.
Compare toxicity | Approximately up to 69 months after randomization of the first patient
  To compare toxicity according to CTCAE v5 between arms
Compare Quality of Life | Approximately up to 69 months after randomization of the first patient
  To compare Quality of Life between arms via validated questionnaires such as QLQ-C30, MY20, EQ-5D-5L
Compare relative dose intensity | Approximately up to 69 months after randomization of the first patient
  To compare relative dose intensity (RDI) of daratumumab, lenalidomide and dexamethasone between arms.

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Zweegman, Prof Dr MD, Principal Investigator — Amsterdam UMC
Locations (38):
- Netherlands (38):
  - NL-Den Bosch-JBZ, 's-Hertogenbosch
  - NL-Almere-FLEVOZIEKENHUIS, Almere Stad
  - NL-Amersfoort-MEANDERMC, Amersfoort
  - NL-Amsterdam- UMC, Amsterdam
  - NL-Amsterdam-AmsterdamUMC, Amsterdam
  - NL-Apeldoorn-GELREAPELDOORN, Apeldoorn
  - NL-Arnhem-RIJNSTATE, Arnhem
  - NL-Assen-WZA, Assen
  - NL-Beverwijk-RKZ, Beverwijk
  - NL-Delft-RDGG, Delft
  - NL-Deventer-DZ, Deventer
  - NL-Dordrecht-ASZ, Dordrecht
  - Nij Smellinghe Ziekenhuis, Drachten
  - NL-Ede-ZGV, Ede
  - NL-Emmen-SCHEPER, Emmen
  - NL-Enschede-MST, Enschede
  - NL-Goes-ADRZ, Goes
  - NL-Gorinchem-BEATRIX, Gorinchem
  - NL-Groningen-MARTINI, Groningen
  - NL-Hardenberg-SAXENBURGH, Hardenberg
  - NL-Harderwijk-STJANSDALHARDERWIJK, Harderwijk
  - NL-Helmond-ELKERLIEK, Helmond
  - NL-Hilversum-TERGOOI, Hilversum
  - NL-Hoofddorp-SPAARNEGASTHUIS, Hoofddorp
  - NL-Hoorn-DIJKLANDERHOORN, Hoorn
  - Alrijne Ziekenhuis Leiderdorp, Leiderdorp
  - HMC Antoniushove, Leidschendam
  - NL-Roosendaal-BRAVIS, Roosendaal
  - NL-Rotterdam-IKAZIA, Rotterdam
  - NL-Schiedam-FRANCISCUSVLIETLAND, Schiedam
  - NL-Sittard-Geleen-ZUYDERLAND, Sittard
  - NL-Sneek-ANTONIUSSNEEK, Sneek
  - NL-Terneuzen-ZORGSAAM, Terneuzen
  - NL-Tilburg-ETZ, Tilburg
  - NL-Uden-BERNHOVEN, Uden
  - NL-Venlo-VIECURI, Venlo
  - NL-Zaandam-ZAANSMC, Zaandam
  - NL-Zwolle-ISALA, Zwolle

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: HOVON website — https://hovon.nl/en